CLINICAL TRIAL: NCT02138396
Title: Single-Dose, Open-Label, Two-Period, Two-Treatment, Two-Sequence Crossover Exploratory Bioavailability Study of Subsys® (Fentanyl Sublingual Spray), 400 mcg, and Fentanyl Citrate Injection 2 mL x 0.05 mg/mL (Total Dose 100 mcg) Under Fasted Conditions
Brief Title: Exploratory Bioavailability of Fentanyl Sublingual Spray Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: INS-13-019
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Bioavailability
MeSH Terms: interventions — Fentanyl; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FSS first, then FCI (Experimental): At each of two treatment visits participants fast for 10 hours before dosing, and receive naltrexone before and after dosing. Participants in this group receive a single dose of fentanyl sublingual spray (FSS) at the first visit. After a washout period of at least seven days, they receive a single intramuscular fentanyl citrate injection (FCI) at the second treatment visit.
  Interventions: Drug: Fentanyl Sublingual Spray (FSS); Drug: Fentanyl Citrate Injection (FCI); Drug: Naltrexone
- FCI first, then FSS (Experimental): At each of two treatment visits participants fast for 10 hours before dosing, and receive naltrexone before and after dosing. Participants in this group receive a single intramuscular fentanyl citrate injection (FCI) at the first visit. After a washout period of at least seven days, they receive a single dose of fentanyl sublingual spray (FSS) at the second treatment visit.
  Interventions: Drug: Fentanyl Sublingual Spray (FSS); Drug: Fentanyl Citrate Injection (FCI); Drug: Naltrexone

INTERVENTIONS:
Drug: Fentanyl Sublingual Spray (FSS) — A single dose of fentanyl, 400 mcg per sublingual spray
  Other Names: Subsys®
Drug: Fentanyl Citrate Injection (FCI) — A single dose of fentanyl citrate, 100 mcg per intramuscular injection
Drug: Naltrexone — Naltrexone is provided as a 50 mg tablet before and after product dosing to minimize unacceptable adverse effects of fentanyl.

SUMMARY:
The objective of this study is to compare the rate of absorption and bioavailability of fentanyl sublingual spray 400 mcg to fentanyl citrate 100 mcg by intramuscular injection.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception
* Good access to veins on both sides
* Willing and able to remain confined in the study unit for the entire duration of each treatment period and comply with restrictions related food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Intolerance to venipuncture or injections
* Presence or history of oral disease, irritation or piercings
* Allergy or adverse response to fentanyl, naltrexone, or related drugs
* Tattoos, scarring, or other skin abnormality at planned injection sites
* History or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise: 1) the safety or well-being of the participant or study staff; 2) the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding); 3) the analysis of results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) by mode of administration | within 36 hours after dosing

SECONDARY OUTCOMES:
Area under the concentration-time curve [AUC(last)] by mode of administration | prior to the intial dose, at 5, 10, 20, 30, and 40 minutes postdose, and at 1.0, 1.25, 1.5, 2.0, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, and 36 hours post-dose
Area under the curve extrapolated to infinity [AUC(inf)] by mode of administration | prior to the intial dose, at 5, 10, 20, 30, and 40 minutes postdose, and at 1.0, 1.25, 1.5, 2.0, 4.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, and 36 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: George J Atiee, MD, Principal Investigator — Worldwide Clinical Trials Early Phase Services, LLC
Locations (1):
- Worldwide Clinical Trials Early Phase Services, LLC, San Antonio, Texas, United States